CLINICAL TRIAL: NCT02982915
Title: Effects of Intravenous Delivery of Lomecel-B (Formerly Allogenic Longeveron Human Mesenchymal Stem Cells (LMSCs)) on VaccinE-Specific Antibody Responses in Subjects With Aging Frailty
Brief Title: Lomecel-B on Vaccine-Specific Antibody- Response in Subjects With Aging Frailty
Acronym: HERA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Longeveron Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00-0000-03
Record Dates: First submitted 2016-11-17; First posted 2016-12-06 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Aging Frailty
MeSH Terms: interventions — Influenza Vaccines; Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pilot Phase- Cohort A (Experimental): Single dose of 20 million Longeveron Mesenchymal Stem Cells (LMSCs) will be delivered followed by vaccination with Fluzone High-Dose at 1 week post-infusion.
  Interventions: Biological: Longeveron Mesenchymal Stem Cells (LMSCs); Biological: Fluzone High Dose Vaccine
- Pilot Phase Cohort B & C (Experimental): Single dose of 100 million Longeveron Mesenchymal Stem Cells (LMSCs) followed by vaccination with Fluzone High-Dose at either 1 week (Cohort B) or 4 weeks (Cohort C) post infusion.
  Interventions: Biological: Longeveron Mesenchymal Stem Cells (LMSCs); Biological: Fluzone High Dose Vaccine
- Double-Blind,Randomized,Placebo Phase (Experimental): 2 cohorts to receive a single infusion of 100 million Longeveron Mesenchymal Stem Cells (LMSCs) (Cohort A: 30 subjects) or placebo (Cohort B:30 subjects) followed by vaccination with Fluzone High-Dose.
  Interventions: Biological: Longeveron Mesenchymal Stem Cells (LMSCs); Biological: Fluzone High Dose Vaccine

INTERVENTIONS:
Biological: Longeveron Mesenchymal Stem Cells (LMSCs) — Intravenously delivered
  Other Names: Lomecel-B
Biological: Fluzone High Dose Vaccine — Intramuscular injection

SUMMARY:
This is a phase I/II, randomized, blinded and placebo-controlled study to test the safety and efficacy of Lomecel-B for improving vaccine immune response.

DETAILED DESCRIPTION:
A pilot phase will consist of a 3 subject safety run-in, followed by 20 subject randomized phase to evaluate influenza vaccine response at 1 week and 4 weeks post infusion of Lomecel-B (Formerly LMSCs). This will be followed by a double-blinded, randomized, placebo-controlled phase.

ELIGIBILITY:
Inclusion Criteria:

* be willing and able to provide written informed consent and comply with all procedures required by the protocol.
* be 65 - 90 years of age at the time of signing the Informed Consent Form.
* have a diagnosis of Aging Frailty, with a score of 4 to 7 using the Canadian Frailty Scale.
* have a six-minute walk test (6MWT) distance of 200m - 400m for each of 2 trials, and the 2 trials must be within 15% of each other.
* have total bilirubin between 0.3 - 1.9 mg/dL.

Exclusion Criteria:

* be unwilling or unable to perform any of the assessments required by the Protocol.
* score ≤24 on the Mini Mental State Examination (MMSE).
* have previously received current year's flu-vaccine.
* have any contraindication to receiving a vaccine.
* have a Hemoglobin A1c (HbA1c) level >9.0%.
* be diagnosed with malignancy (subjects without a recurrence in the last 2.5 years will be allowed) except curatively-treated basal cell carcinoma, melanoma in situ, or cervical carcinoma.
* have a condition that projected to limit the life-expectancy to ≤1 year.
* have autoimmune disease (e.g., rheumatoid arthritis).
* be using medication(s) known to alter immune response, e.g., high-dose corticosteroids.
* have HIV, AIDS, or other immunodeficiency.
* test positive for hepatitis B virus

  * If the subject tests positive for anti-HBc or anti-HBs, they must be receiving treatment for Hepatitis B virus prior to infusion and remain on treatment throughout the study.
* test positive for viremic hepatitis C, HIV1, HIV2, or syphilis.
* have a resting blood oxygen saturation of <93% (measured by pulse oximetry).
* be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraception.
* have documented current substance and/or alcohol abuse.
* have known allergies to latex or eggs.
* have a known hypersensitivity to dimethyl sulfoxide (DMSO).
* be an organ transplant recipient (other than corneal, bone, skin, ligament, or tendon transplant).
* be actively listed (or expected to be listed) for transplant of any organ (other than corneal, bone, skin, ligament, or tendon transplant).
* have any clinically important abnormal screening laboratory values, including but not limited to:

  * hemoglobin <10.0 g/dL.
  * white blood cell count < 2500/mm3.
  * platelets < 100,000/mm3.
  * prothrombin time/international normalized ratio (PT/INR) ˃ 1.5 not due to a reversible cause (i.e. Coumadin).
* aspartate transaminase, alanine transaminase, or alkaline phosphatase ˃ 2 times upper limit of normal.
* have a sitting or resting systolic blood pressure >180 mm Hg or diastolic blood pressure >110 mm Hg at Screening.
* have any serious illness or any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the subject or preclude successful completion of the study, or that may compromise the validity of the study.
* be currently participating in an investigational therapeutic or device trial, or have participated in an investigational therapeutic or device trial within the previous 30 days, or participate in any other clinical trial for the duration of the time that the subject actively participates in this trial.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
The incidence of any treatment-emergent serious adverse event (TE-SAE), defined as one or more of the following untoward medical occurrences within 30 days after infusion as assessed by the following: | 30 days after infusion
  * Is life-threatening (e.g., stroke or non-fatal pulmonary embolism).
  * Requires inpatient hospitalization or prolongation of existing hospitalization.
  * Results in persistent or significant disability/incapacity.
  * Results in death
  * Results in other clinically significant untoward laboratory test result(s) or medical condition(s), determined per Investigator's judgment.
The ability of Lomecel-B (LMSC) treatment to improve inactivation of influenza virus as assessed by validated hemagglutination inhibition (HAI) assays. | Baseline Visit, Vaccination Visits, Weeks 1, 2, 4, Month 6 and Month 12 Follow-Up Visits.
  Measurements of validated hemagglutination inhibition (HAI) assays at follow up visits.

SECONDARY OUTCOMES:
Changes from baseline between the LMSC and placebo cohorts as assessed by plasma cytokine levels: | Baseline, month 6 and month 12 after infusion
  Plasma levels of interleukins measured in pg/mL.
Differences in rate of decline from Aging Frailty | Baseline, month 6 and month 12 after infusion
  Change in Clinical Frailty rating
Assessed by the Falls Efficacy Scale-International and Performance Oriented Mobility Assessment | Baseline, month 6 and month 12 after infusion
  Change in risk of falling
PROMIS Short Form 20a questionnaire | Baseline, month 6 and month 12 after infusion
  Change in subject quality of life as assessed by participant-reported outcomes.
PROMIS Mobility questionnaire | Baseline, month 6 and month 12 after infusion
  Change in subject quality of life as assessed by participant-reported outcomes.
PROMIS Upper Extremity questionnaire | Baseline, month 6 and month 12 after infusion
  Change in subject quality of life as assessed by participant-reported outcomes.
Short Form 36 questionnaire | Baseline, month 6 and month 12 after infusion
  Change in subject quality of life as assessed by participant-reported outcomes.
IIEF questionnaire | Baseline, month 6 and month 12 after infusion
  Change in subject quality of life as assessed by participant-reported outcomes.
SQOL-F questionnaire | Baseline, month 6 and month 12 after infusion
  Change in subject quality of life as assessed by participant-reported outcomes.
Death from any cause | Within 12 months after infusion
  Number of participants that die from any cause while enrolled on the trial and after being treated with LMSCs.
Falls Efficacy Scale-International (FES-I) | Baseline, month 6 and month 12 after infusion
  Change by participant-reported outcomes. Minimum 16 (no concern about falling) to maximum 64 (severe concern about falling)
Changes from baseline between the LMSC and placebo cohorts as assessed by B & T cell levels: | Baseline, month 6 and month 12 after infusion
  Plasma levels of B & T Cells.
Rate of decline in Aging Frailty status as assessed by the 6 minute walk test | Baseline, month 6 and month 12 after infusion
  Distance in meters walked in 6 minutes
Rate of decline in Aging Frailty status as assessed by the Short Physical Performance Battery (SPPB) | Baseline, month 6 and month 12 after infusion
  Short Physical Performance Battery Assessment
Rate of decline in Aging Frailty status as assessed by the Tinetti POMA Test | Baseline, month 6 and month 12 after infusion
  TInetti POMA assessment
Rate of decline in Aging Frailty status as assessed by the Weight Loss | Baseline, month 6 and month 12 after infusion
  Weigh measurements at visits
Rate of decline in Aging Frailty status as assessed by the Handgrip Test | Baseline, month 6 and month 12 after infusion
  Handgrip strength via dynamometer.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Clinical Research of South Florida, Coral Gables, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - University of Miami, Miami, Florida
  - Vista Health Research, Miami, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Optimal Research LLC, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: No